CLINICAL TRIAL: NCT01818089
Title: Monitoring of Lung Sounds of Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-116
Record Dates: First submitted 2013-02-15; First posted 2013-03-26 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung Sound Analyzer: Patient with pneumonia admitted to hospital will receive additional auscultation with lung sound analyzing stethoscope
  Interventions: Device: Lung sound analyzer

INTERVENTIONS:
Device: Lung sound analyzer — Patients will be aucultated with lung sound analyzer. The auscultation will be done three times daily during the duration of the complete hospital stay.
  Other Names: Electronic stethoscope; Model 3200; Littmann 3M

SUMMARY:
The aim of this study is to investigate if any correlation between lung sounds of pneumonia patients and the clinical development or therapy of the pneumonia exists.

ELIGIBILITY:
Inclusion Criteria:

* ambulant aquired pneumonia with typically radiological signs
* hospitalisation at medical clinic I, university hospital Aachen
* age at least > 18 years
* CRB-65 score > 1
* CRP> 60mg/l
* fever
* lung sounds audible by stethoscope
* legal capacity and being able to understand and to follow the instructions of the study staff
* being able to consent and being able to understand the importance and the consequence of the study
* not being accomondated in an institution

Exclusion Criteria:

* pneumonia acquired in a hospital
* artificial respiration or other means for supporting respiration
* allergic reaction because of skin contact with polymers
* pregnancy or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ambulant aquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Sound of lungs | 5 days
  3 times a day for longest 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Cornelissen, MD, Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany